CLINICAL TRIAL: NCT04303845
Title: Erenumab For Treatment of Hemicrania Continua
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: difficulty with recruitment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rashmi B. Halker Singh MD, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-007088
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Results first posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-01

CONDITIONS: Hemicrania Continua
MeSH Terms: interventions — erenumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with Erenumab (Experimental): Subjects diagnosed with hemicrania continua will receive single dose of Erenumab
  Interventions: Drug: Erenumab

INTERVENTIONS:
Drug: Erenumab — 140 mg of erenumab via subcutaneous injection

SUMMARY:
This research is being conducting to learn if the study drug erenumab is successful in treating hemicrania continua. The study is also evaluating the safety and tolerability of erenumab in individuals being treated for hemicrania continua.

ELIGIBILITY:
Inclusion Criteria

* Adults over the age of 18-66
* At least a 12 month history of hemicrania continua (unremitting subtype) according to International Classification of Headache Disorders, 3rd Edition (ICHD-3)1
* Previous or current complete response to indomethacin
* Stable preventive treatment for at least 2 months and no anticipated need to adjust/add current headache prevention treatment

Exclusion Criteria

* Nonresponse to a therapeutic dose of indomethacin for hemicrania continua when used for at least 1 week
* Pregnant or lactating subjects
* Use of barbiturate or opioid >6 days per month; history of chronic migraine
* History of previous trigeminal-autonomic cephalalgia
* History within previous 2 months of interventional procedure for headache (occipital or other extracranial nerve block, sphenopalatine ganglion block, cervical facet block, facet rhizotomy)
* History of cranial nerve/rhizolysis
* Botulinumtoxin injection with previous 4 months
* Parenteral infusion of or oral corticosteroid use for more than 3 days within 4 weeks prior to screening phase

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Halker Singh, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment With Erenumab: Subjects diagnosed with hemicrania continua received single dose of Erenumab
  Erenumab: 140 mg of erenumab via subcutaneous injection
Period: Overall Study
Arm/Group | Treatment With Erenumab
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment With Erenumab
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (19.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Headache Days
Description: The total number of days per month (28 days) with headache of any kind/severity
Time Frame: 4 weeks post erenumab treatment
Population: Terminated study due to low enrollment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment With Erenumab
Number analyzed (Participants) | 2
days | 24.5 (4.9)

2. Secondary Outcome: Migraine Days
Description: Total number of days per month (28 days) with migraines
Time Frame: 4 weeks post erenumab treatment
Population: Terminated study due to low enrollment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment With Erenumab
Number analyzed (Participants) | 2
days | 0.5 (0.7)

3. Secondary Outcome: Headache Freedom
Description: Total number of days per month (28 days) with complete headache freedom
Time Frame: 4 weeks post erenumab treatment
Population: Terminated study due to low enrollment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment With Erenumab
Number analyzed (Participants) | 2
days | 3.5 (4.9)

4. Secondary Outcome: Remission Rate
Description: Number of participants who do not have any occurrence of headache
Time Frame: 4 weeks post erenumab treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Erenumab
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 8 weeks.
Arm/Group | Treatment With Erenumab
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Erenumab (N=2)
Worsening of pre-existing medical condition (General disorders) | 1

LIMITATIONS AND CAVEATS:
Terminated study due to low enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT04303845/Prot_SAP_000.pdf